CLINICAL TRIAL: NCT06637813
Title: Establishment of a Database of HIV Subjects Initiating or Simplifying Dual Therapy With Dolutegravir/Lamivudine
Acronym: NEW_ODOACRE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7059
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: HIV -1 Infection
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood biospecimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Blood sampling for evaluation of biomarkers — Non-routine diagnostic test evaluations

SUMMARY:
The introduction of combination antiretroviral therapy (cART) has completely revolutionized the management of HIV-positive patients, drastically reducing HIV-associated mortality and morbidity. In fact, the course of HIV infection has transformed into a chronic disease. The availability of different classes of antiretroviral drugs, such as nucleoside and non-nucleoside reverse transcriptase inhibitors (NRTIs, NNRTIs), protease inhibitors (PIs), integrase inhibitors (INSTIs) and viral entry inhibitors (IEs) that act in different phases of the HIV life cycle, together with careful patient management, has allowed us to obtain long-lasting therapeutic efficacy in the vast majority of Italian patients, making this infection a chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* patients treated with triple therapy who simplify to 3TC+DTG
* patients treatment-naive who start a dual therapy with 3TC+DTG from clinical practice

Exclusion Criteria:

* lack of willingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV subjects treated with Dovato from 2015 to 2022. (retrospective cohort) or who will start treatment from clinical practice with Dovato
Sampling Method: Non-Probability Sample
Enrollment: 1220 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2034-10-30 (Estimated)

PRIMARY OUTCOMES:
Establishment of a database | 10 years
  Systematic and continuous collection of data related to clinical, laboratory and treatment characteristics of patients who simplify from triple standard ART or who continue dual therapy with 3TC+DTG, or treatment-naive patients who start the dual regimen with 3TC+DTG. The data will be useful for the evaluation of diagnostic and multiparametric algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Di Giambenedetto, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: Undecided